CLINICAL TRIAL: NCT03478150
Title: Evaluation of The Antibacterial Effect of Laser Diode and Zinc Oxide Nano-particles on Streptococcus Mutans Bacteria Used as Cavity Disinfectants in Deep Carious Lesions : A Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Antibacterial Effect of Laser Diode and Zinc Oxide Nano Particles in Cavity Disinfection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Atef Khattab, master student at the department of conservative and aesthetic dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: oper151
Record Dates: First submitted 2018-03-18; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the examiner who will carry the microbiological analysis of dentin samples will be blinded to the type of agent applied during treatment. Finally, the treatment results will be assessed blindly by a statistician.
  Blinding:
  Blinding of the operator is not possible, because the natures of both interventions are obviously different. The operator is blinded until randomization into groups, to avoid biases with regard to the application of antibacterial agent. Also, the examiner who will carry the microbiological analysis of dentin samples will be blinded to the type of agent applied during treatment. Finally, the treatment results will be assessed blindly by a statistician also to avoid the risk of bias of results in favor of one intervention over the other.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- zinc oxide nano-particles (Experimental): The zinc oxide nano-powder will be mixed with ethanol and applied in the cavity, where the ethanol evaporates, while the zinc oxide nano-particles infiltrate into the carious floor of the cavity.
  Interventions: Other: zinc oxide nano-particles
- laser diode (Experimental): Each cavity will be irradiated in contact mode with continuous wave of radiation. The laser light is transferred through a 600µm flexible fiber optic tip by a special hand piece. The fiber optic will be disinfected for each use by 70% ethyl alcohol and inserted inside the cavity to 1mm with a spiral continuous movement clockwise from the top to the floor and anti-clockwise in the reverse direction. This procedure improves the distribution of the laser light inside the cavity and to avoid excessive heat generation in the internal cavity surface. Irradiation time will be 15 seconds and repeated 5 times with 15 second intervals with contact, according to manufacture instructions. During this study the output power will be adjusted at 1.5W.
  Interventions: Device: laser diode

INTERVENTIONS:
Other: zinc oxide nano-particles — The zinc oxide nano-powder will be mixed with ethanol
  Arms: zinc oxide nano-particles
Device: laser diode — The laser light is transferred through a 600µm flexible fiber optic tip by a special hand piece. the output power will be adjusted at 1.5W.
  Arms: laser diode

SUMMARY:
this is a randomized controlled clinical trial, evaluating the antibacterial effect of laser diode and zinc oxide nano-particles when used as cavity disinfectants.Two groups, including 15 patients each, will be randomly allocated so that each group receives one of either interventions (15 patients will undergo cavity disinfection by laser diode, while the other 15 patients will undergo cavity disinfection by zinc oxide nano-particles). For each patient, a dentin sample will be taken before and after cavity disinfection. The dentin samples will be microbiologically analyzed to assess the difference in the bacterial count (out come assessment). The results will be statistically analyzed.

DETAILED DESCRIPTION:
This study will be carried out on adult patients attending to the department of conservative dentistry at The Faculty of Oral and Dental Medicine, Cairo University, Egypt. The procedures will be carried out by postgraduate student Sarah Atef Khattab (B.D.S. 2011) from Cairo university without an assistant. The researcher will bear ultimate responsibility for all activities associated with the conduct of a research project including recruitment of patients, explaining and performing the procedures to them.

A : Excavation protocol:

The teeth of the patients that meet inclusion criteria will be anaesthetized, isolated with a rubber dam. Cavity opened using conventional high-speed rotary instruments. The central cariogenic biomass and the superficial parts of the necrotic dentine will be removed with round burs. Caries lesion will be completely removed in the enamel/dentin junction. The excavation procedure will be terminated as soon as the soft and wet dentine was removed and the remaining tissue was leathery but not hard on exploring. A dentinal sample will then be collected from the base of the cavity using sterile spoon excavator as a baseline for bacteriological assessment. Then, after application of either interventions , another dentinal sample will be collected using a sterile excavator and transferred into sterile tubes and transferred to the laboratory for microbiological analysis.

b. Application of the interventions: b.1: laser diode Each cavity will be irradiated in contact mode with continuous wave of radiation. The laser light is transferred through a 600µm flexible fiber optic tip by a special hand piece. The fiber optic will be disinfected for each use by 70% ethyl alcohol and inserted inside the cavity to 1 millimeter with a spiral continuous movement clockwise from the top to the floor and anti-clockwise in the reverse direction. This procedure improves the distribution of the laser light inside the cavity and to avoid excessive heat generation in the internal cavity surface. Irradiation time will be 15 seconds and repeated 5 times with 15 second intervals with contact, according to manufacture instructions. During this study the output power will be adjusted at 1.5 Watt.

b.2: Zinc oxide nano-particles: The zinc oxide nano-powder will be mixed with ethanol and applied in the cavity, where the ethanol evaporates, while the zinc oxide nano-particles infiltrate into the carious floor of the cavity.

N.B: In both methods, a dentin sample will be taken before the application of the disinfectant, then the zinc oxide nano-particles are applied in the cavity and left for 5 minutes, then another sample will be taken. The second specimen will be compared to the first specimen taken before cavity disinfection, regarding the streptococcus mutans count.

c .Assessment of Outcome: Samples of carious dentin will be collected with sterile excavator before and after application of both interventions. The dentin samples will be transferred to sterile container containing a 1millilitre thioglycollate medium used as a carrier, then this sterile container will be kept in an ice box and taken to the microbiology laboratory for processing, within an hour, by another examiner who is blinded to the type of agent applied after partial caries removal. Samples will be vortexed for two minutes, decimally diluted and 0.1 ml will be plated on Mitis Salivarius Bacitracin agar plates, these plates will be incubated anaerobically for 48 hour at 37 degree celcius then aerobically for 24 hour at room temperature. The number of colonies will be expressed as colony-forming units (CFU/ml) compared before and after application of the antibacterial agent.

ELIGIBILITY:
Inclusion Criteria:

* Normal adults will be recruited in this study, with free medical history
* Have not received antibiotic therapy since 1 month before sampling
* Good oral hygiene
* Co-operative patients approving the trial
* In each patient required one or two deeply carious class v cavities either upper or lower permanent anterior teeth

Exclusion Criteria:

* Subjects with a history of allergy to any of the drugs or chemicals used in the study
* History of pulp pathology of the teeth which indicates root canal treatment is not included in the study
* Pregnancy and Lactating mothers
* Patients with any systematic problems or mental or physical disability
* Heavy smoking
* Xerostomia
* Lack of compliance

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in the bacterial Count (Streptococcus Mutans) CFU/ml after cavity disinfection | About one year
  Samples of carious dentine will be collected with sterile excavator before and after application of both interventions. The dentine samples will be transferred to sterile container containing a 1mL thioglycollate medium used as a carrier, then this sterile container will be kept in an ice box and taken to the microbiology laboratory for processing, within an hour, by another examiner who is blinded to the type of agent applied after partial caries removal. Samples will be vortexed for two minutes, decimally diluted and 0.1 ml will be plated on Mitis Salivarius Bacitracin agar plates, these plates will be incubated anaerobically for 48 hour at 37ºC then aerobically for 24 hour at room temperature. The number of colonies will be expressed as colony-forming units (CFU/ml) compared before and after application of the antibacterial agent.

CONTACTS AND LOCATIONS:
Overall Officials: Mona I Riad, professor, Study Chair — Cairo University; Rasha Raafat, lecturer, Study Director — Cairo University
Locations (1):
- sarah Atef khattab, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohan PV, Uloopi KS, Vinay C, Rao RC. In vivo comparison of cavity disinfection efficacy with APF gel, Propolis, Diode Laser, and 2% chlorhexidine in primary teeth. Contemp Clin Dent. 2016 Jan-Mar;7(1):45-50. doi: 10.4103/0976-237X.177110. PMID 27041900